CLINICAL TRIAL: NCT02910206
Title: Comparative Effect of Etomidate and Propofol on Major Complications After Abdominal Surgery in Elderly Patients
Brief Title: Etomidate to Improve Outcome in Elderly Patients
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, Dr., Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJH-A-2015-12-01
Record Dates: First submitted 2016-06-30; First posted 2016-09-21 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Complications
Keywords: etomidate; propofol
MeSH Terms: conditions — Postoperative Complications | interventions — Etomidate; Propofol; Sufentanil; cisatracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: participants were anesthetized and were unaware of the grouping. Care providers did not know the grouping. Specific investigators who did the intervention were aware of the grouping. The outcome assessors and the data analyzers did not know the grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- etomidate (Experimental): etomidate is given for maintenance of general anesthesia,combined with sufentanil and cisatracurium
  Interventions: Drug: Etomidate; Drug: Sufentanil; Drug: Cisatracurium
- propofol (Experimental): propofol is given for maintenance of general anesthesia,combined with sufentanil and cisatracurium
  Interventions: Drug: propofol; Drug: Sufentanil; Drug: Cisatracurium

INTERVENTIONS:
Drug: Etomidate — etomidate is given intravenously
  Arms: etomidate
Drug: propofol — propofol is given intravenously
  Arms: propofol
Drug: Sufentanil — sufentanil is given intravenously
Drug: Cisatracurium — Cisatracurium is given intravenously

SUMMARY:
Elderly patients have high mortality and postoperative complications rate after surgery, especially postoperative cardiac complications. A meta-analysis revealed haemodynamic intraoperative events significantly increased the risk of postoperative cardiac complications.To limit the risk, optimize the intraoperative management of circulation is essential. Anesthetic drug may effect on the haemodynamic intraoperative, reduction of postoperative complications should aimed at choosing the optimal anesthetic drug with minimal effect on haemodynamic.So this study is to explore the comparative efficacy and safety of anesthetic drug (etomidate or propofol) in elderly patients

ELIGIBILITY:
Inclusion Criteria:

* Aged between 65 and 80 years old.
* Patients scheduled for elective gastrointestinal surgery under general anesthesia.

Exclusion Criteria:

* Expected duration of surgery < 1 or >4 hours
* American Society of Anesthesiologists status >III
* Body Mass Index < 18 kg/m2 or> 25 kg/m2
* Cerebrovascular accident occurred within the previous 3 months,such as stroke or transient ischemic attack
* Unstable angina and myocardial infarction occurred within the previous 3 months
* Patients with serious hepatic dysfunction ( the serum level of alanine transaminase, conjugated bilirubin, aspartate transaminase, alkaline phosphatase or total bilirubin is 2 folds more than upper normal limit) or renal dysfunction(creatinine clearance rate less than 30 milliliter per minute).
* Diabetic patients with complication (diabetic ketoacidosis, hyperosmotic coma,all kinds of infection, macroangiopathy, diabetic nephropathy, retinopathy, diabetic cardiomyopathy, diabetic neuropathy, diabetic foot).
* Preoperative blood pressure more than or equal to 180/110 mmHg
* Confirmed or suspected of narcotic analgesics abusing or long term using
* Taking corticosteroids or immunosuppressive agents for more than 10 days with the previous 6 months or had history of adrenal suppression or immune system disease.
* Patients with thyroid hypofunction.
* Patients with history of asthma.
* Patients with history of surgery within previous 3 months.
* Patients allergic or contraindicated to propofol or etomidate
* Patients participated in other study within the last 30 days

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1917 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with complications defined by ICD (International codes of diseases)-9 | From the moment of giving sufentanil to the moment of discharge from hospital,up to 7 days

SECONDARY OUTCOMES:
the time to awake from anesthesia | From stopping etomidate or propofol infusion to awake, approximately 30 minutes
the time to withdraw tracheal tube from anesthesia | From end of etomidate or propofol infusion to recovery of spontaneous breathing and withdrawal of tracheal tube,approximately 30 minutes
the time to discharge from post-anesthesia care unit | From admit into post-anesthesia care unit to discharge from post-anesthesia care unit,on an average of 30 minutes
the time to discharge from hospital | From end of surgery to discharge from hospital,on an average of 7 days
Post Operative Nausea And vomiting score | 6 hours, 24 hours, 48 hours and 72 hours after end of surgery，approximately 6 hours, 24 hours, 48 hours and 72 hours respectively
  score:0,no nausea and vomiting; 1,nausea without vomiting; 2,vomiting
pain on visual analogue scale | 6 hours after end of surgery，approximately 6 hours
satisfaction on visual analogue scale by the patients | 24 hours after end of surgery
  patients will be asked to score their satisfaction on anesthesia on a visual analogue, 0 is for extremely unsatisfied, 10 is for totally satisfied
comfort on visual analogue scale by the patients | 24 hours after end of surgery
  patients will be asked to score their comfort during and after anesthesia on a visual analogue, 0 is for extremely unsatisfied, 10 is for totally satisfied
incidence of hypotension during anesthesia | from start of surgery to end of surgery, on an average of 2.5 hours
  hypotension is defined as decrease of systemic blood pressure more than 20% of baseline
incidence of hypertension during anesthesia | from start of surgery to end of surgery, on an average of 2.5 hours
  hypotension is defined as increase of systemic blood pressure more than 20% of baseline
percentage of patients needed vasoactive agents during anesthesia | from start of surgery to end of surgery, on an average of 2.5 hours
concentration of serum Cortisol by radioimmunoassay | 24hours,48hours and 72hours after extubation，approximately 24 hour, 48 hour and 72 hour respectively
concentration of serum aldosterone by radioimmunoassay | 24hours,48hours and 72hours after extubation，approximately 24 hour, 48 hour and 72 hour respectively
concentration of serum Adrenocorticotropichormone(ACTH) by radioimmunoassay | 24hours,48hours and 72hours after extubation，approximately 24 hour, 48 hour and 72 hour respectively
death by 6 months after surgery | from end of surgery to 6 months after surgery
death by 12 months after surgery | from end of surgery to 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lize Xiong, PhD, Study Chair — Xijing hosptial
Locations (1):
- Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Du Y, Chen YJ, He B, Wang YW. The Effects of Single-Dose Etomidate Versus Propofol on Cortisol Levels in Pediatric Patients Undergoing Urologic Surgery: A Randomized Controlled Trial. Anesth Analg. 2015 Dec;121(6):1580-5. doi: 10.1213/ANE.0000000000000981. PMID 26496368
- [Background] Aghdaii N, Ziyaeifard M, Faritus SZ, Azarfarin R. Hemodynamic Responses to Two Different Anesthesia Regimens in Compromised Left Ventricular Function Patients Undergoing Coronary Artery Bypass Graft Surgery: Etomidate-Midazolam Versus Propofol-Ketamine. Anesth Pain Med. 2015 Jun 22;5(3):e27966. doi: 10.5812/aapm.27966v2. eCollection 2015 Jun. PMID 26161330
- [Background] Song JC, Lu ZJ, Jiao YF, Yang B, Gao H, Zhang J, Yu WF. Etomidate Anesthesia during ERCP Caused More Stable Haemodynamic Responses Compared with Propofol: A Randomized Clinical Trial. Int J Med Sci. 2015 Jul 3;12(7):559-65. doi: 10.7150/ijms.11521. eCollection 2015. PMID 26180512
- [Background] Kaushal RP, Vatal A, Pathak R. Effect of etomidate and propofol induction on hemodynamic and endocrine response in patients undergoing coronary artery bypass grafting/mitral valve and aortic valve replacement surgery on cardiopulmonary bypass. Ann Card Anaesth. 2015 Apr-Jun;18(2):172-8. doi: 10.4103/0971-9784.154470. PMID 25849685
- [Derived] Lu Z, Zheng H, Chen Z, Xu S, Chen S, Mi W, Wang T, Chai X, Guo Q, Zhou H, Yu Y, Zheng X, Zhang J, Ai Y, Yu B, Bao H, Zheng H, Huang W, Wu A, Deng X, Ma H, Ma W, Tao L, Yang X, Zhang J, Liu T, Ma HP, Liang W, Wang X, Zhang Y, Du W, Ma T, Xie Y, Xie Y, Li N, Yang Y, Zheng T, Zhang C, Zhao Y, Dong R, Zhang C, Zhang G, Liu K, Wu Y, Fan X, Tan W, Li N, Dong H, Xiong L. Effect of Etomidate vs Propofol for Total Intravenous Anesthesia on Major Postoperative Complications in Older Patients: A Randomized Clinical Trial. JAMA Surg. 2022 Oct 1;157(10):888-895. doi: 10.1001/jamasurg.2022.3338. PMID 35947398